CLINICAL TRIAL: NCT03838432
Title: The Efficacy and Safety of Composite Steep-pulse(High-frequency Irreversible Electroporation) Treatment Apparatus Used in Prostate Cancer Ablation Therapy : a Multicenter, Single-arm, Objective Performance Criteria Trial
Brief Title: The Composite Steep-pulse Treatment Apparatus Used in Prostate Cancer Ablation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Military Medical University (Other)
Collaborators: RenJi Hospital (Other); Peking Union Medical College Hospital (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, yinghao Sun, director, head of uroglogy department, clinical professor, Second Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZLC-12-1
Record Dates: First submitted 2018-10-18; First posted 2019-02-12 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: focal therapy; IRE; Composite Steep-pulse Treatment Apparatus; prostate cancer; Multi-center
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Steep Pulse Device (Experimental): Applying the steep pulse to treat the patients with Prostate cancer
  Interventions: Device: Steep Pulse Device

INTERVENTIONS:
Device: Steep Pulse Device — Applying the steep pulse to treat the patients with Prostate cancer

SUMMARY:
This trial is studying the effects and safety in treating patients from five different centers with local prostate cancer, employing Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Apparatus. This device could cause cell irreversible electroporation, which leading necrosis of tumor cells. It also has the ability to prevent nerve,vessel, urethral and capsule unnecessary injury beside the ablation area. Composite Steep-pulse Treatment Apparatus will be used in patients who pass inclusion/exclusion criteria. Safety, quality of life, and histopathological analysis of prostate speciem will be evaluated in each study patients.

DETAILED DESCRIPTION:
Background:

Prostate cancer is the most common cancer in elderly males in western country. It is also a major health concern, especially in China with its greater proportion of elderly men in the general population. Currently, radical prostatectomy(RP) is the mainstream treatment for localized PCa to show a benefit for cancer-specific survival (CSS). However, the patient who underwent RP might suffer from the complication of erectile dysfunction or urinary incontinence. In 2004, a new method using steep pulses to treat tumor was appeared. It showed that steep pulses could bring about Irreversible Electroporation (IRE) of cell, leading tonecrosis of tumor cells. And it seemed to do no harms to the nerve and Vascular epithelial cell. The device of steep pulse had already been approved by FDA in 2011.However, this device of steep pulse has disadvantages like: (1)sever muscle contraction;(2)Urethral injury; (3)Capsule injury;(4)Nerve degeneration. This new device which is called Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Apparatus, may have the potential to conquer these disadvantages.

Purpose:

1. This study will assess the efficacy of Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Apparatus in the treatment of PCa.
2. This study will assess the safety of Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Apparatus in the treatment of PCa.

Methods:

1. patients recruitment
2. transperineal maping prostate biopsy(>20 needle) guided by transrectal ultrasound(TRUS).
3. Irreversible Electroporation of malignant Tumor Cell under Composite Steep-pulse Treatment for the patients with positive biopsy;
4. Some factors such as prostate MRI,the maping prostate biopsy(>20 needle),the histopathological outcomes analysis ect. will be performed to evaluate the efficacy of the treatment.
5. Other factors such as the routine blood test, the routine urine test, the urinary continence ect. will be performed to evaluate the safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The therapy must be thoroughtly understood with the agreement signed
2. Prostate MRI can identify negative extracapsular extension and seminal vesicle involvement,and no evidence of lymphatic metastasis
3. Patients must have confirmed prostate cancer by prostate maping biopsy
4. Low-risk or intermediate risk prostate cancer(PSA<20ng/ml,T1a-T2c,Gleason Score≤7)
5. There must be no evidence of metastatic disease as confirmed by ECT and whole-body MRI
6. No prostatic calculus or prostatic calculus≤5mm
7. Age ≥ 40 - ≤ 85 years
8. Life expectancy of greater than 5 years(WHO Performance Status 0-1)
9. Patients with fertility are willing to take contraceptive measures until the end of the trial

Exclusion Criteria:

1. Patients have previously undergone radical prostatectomy, hormonal therapy or radiotherapy.
2. Patients underwent other surgery before less than 3 months.
3. Patients required long-term medication with anticoagulans or stop taking anticoagulans less than 1 months
4. Patients with clinically significant cardiovascular disease or other serious diseases
5. Patients with metal implants in their bodys(for example,cardiac pacemaker ) and/or with metal implants which located in the range from the first lumbar vertebra(L1) to the middle of femurs.
6. Patients with history of epilepsy
7. Patients with other malignant tumor or patients with hiv.
8. Patients with other serious systemic diseases that the study believes may interfere with the treatment, evaluation, and compliance of the trial;
9. Patients with participation in another clinical trial less than 3 months.
10. Patients with the judge that they are not suitable for this clinical trial

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-01-18 (Estimated)

PRIMARY OUTCOMES:
The result of prostate maping biopsy | 6 Months
  evaluation of pathological analysis from the biopsy sample to confirm if there remain clinically significant prostate cancer
The result of prostate MRI | 6 Months
  evaluation of ablation range from prostate MRI to confirm if there remain suspicious lesions

SECONDARY OUTCOMES:
urinary incontinence | 6 Months
  The rate of urinary incontinence
urination function(IPSS scoring) | 6 Months
  evaluation of urination function by IPSS scoring
sexual function (IIEF-5 scoring) | 6 Months
  evaluation of sexual function by IIEF-5 scoring
urinary catheter retention time | 6 Months
  Record of urinary catheter retention time

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital,Second Military Medical University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang H, Xue W, Yan W, Yin L, Dong B, He B, Yu Y, Shi W, Zhou Z, Lin H, Zhou Y, Wang Y, Shi Z, Ren S, Gao X, Wang L, Xu C. Extended Focal Ablation of Localized Prostate Cancer With High-Frequency Irreversible Electroporation: A Nonrandomized Controlled Trial. JAMA Surg. 2022 Aug 1;157(8):693-700. doi: 10.1001/jamasurg.2022.2230. PMID 35793110
- [Derived] He BM, Xue W, Yan WG, Yin L, Dong BJ, Zhou ZE, Lin HZ, Zhou Y, Wang YQ, Shi ZK, Zhou H, Wang SD, Ren SC, Gao X, Wang LH, Xu CL, Wang HF. A Multicenter Single-Arm Objective Performance Criteria Trial to Determine the Efficacy and Safety of High-Frequency Irreversible Electroporation as Primary Treatment for Localized Prostate Cancer: A Study Protocol. Front Oncol. 2021 Nov 10;11:760003. doi: 10.3389/fonc.2021.760003. eCollection 2021. PMID 34858837